CLINICAL TRIAL: NCT04930406
Title: Impact of Physical Therapy Intervention on Foot and Ankle Function in Children and Adolescents With Non-CNS Cancers
Brief Title: Impact of Physical Therapy Intervention on Foot and Ankle Function
Status: Recruiting | Type: Observational
Sponsor: Children's Hospitals and Clinics of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 1210-108
Record Dates: First submitted 2021-04-27; First posted 2021-06-18 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Neoplasms; Physical Therapy Modalities; Survivorship
MeSH Terms: conditions — Neoplasms | interventions — Physical Therapy Modalities

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Historical control group
- Intervention group
  Interventions: Other: Physical therapy

INTERVENTIONS:
Other: Physical therapy — Had to receive 10 or more visits of physical therapy during the cancer treatment period to qualify for intervention group.
  Groups: Intervention group

SUMMARY:
This research study will investigate the effect of physical therapy intervention on the function of the foot and ankle in children and adolescents with cancer not involving the brain or spinal cord. Children undergoing treatment for cancer can suffer from decreased flexibility, strength, balance and endurance from the cancer and from direct effects of the chemotherapy agents. These deficits have been shown to continue years after treatment end with adult survivors of cancer being less physically active then their siblings. Children, whose chemotherapy includes neurotoxic agents such as vincristine, can develop damage to their peripheral nervous system affecting the strength, sensation, and flexibility in their hands and feet. This can then lead to a change in their walking pattern and likely contributes to decreased physical activity level and fatigue. The principal investigator is currently involved in research with Dr. Laura Gilchrist and Dr. Mary C. Hooke establishing the reliability and validity of a measurement tool to quantify peripheral neuropathy, identifying physical impairments of children with cancer during treatment, and comparing physical performance in children after treatment completion with and without physical therapy intervention. The principal investigator is also completing data analysis on a pilot study investigating the use of ankle foot orthotics in children and adolescents with non-CNS cancer. In this study, the investigators will further the research by measuring the effect of physical therapy intervention on measurements involving the function and structure of the ankle and foot. The investigators will compare participants who have and have not received physical therapy intervention during cancer treatment by administering measurements detailing the function of the foot and ankle in order to further evaluate the benefit of physical therapy for children with cancer. Physical therapy intervention involving children and adolescents with cancer focuses on minimizing the physical impairments caused by chemotherapy and radiation treatment, as well as promoting normal development of motor skills typically obtained by a child in their age group. In the oncology population, physical therapy often targets the foot and ankle as this is most affected by peripheral neuropathy. Interventions include strengthening, balance training, stretching, and orthotic use to allow normal motor skills. Families are instructed in exercises that can be completed at home to further improve their function. This study will examine the difference in the function of the foot and ankle years after intervention in participants who have and have not received these interventions. The investigators will measure neuropathy, ankle flexibility, ankle strength, foot posture, gait mechanics, and endurance in order to fully examine the foot and ankle as well as evaluate relationships between the variables in long-term survivors of pediatric cancer.

ELIGIBILITY:
Inclusion Criteria:

* Historical control group

  * Children and adolescents age 7-30
  * English speaking family
  * Diagnosed with a non-CNS cancer diagnosis with chemotherapy regimen including vincristine, carboplatin, or cisplatin
  * Completed cancer treatment greater than 5 years ago
  * Received less than 2 intervention visits of outpatient physical therapy during cancer treatment

    -• Intervention group
  * Children and adolescents age 7-30
  * English speaking family
  * Completed cancer treatment greater than 5 years ago
  * Greater than 10 physical therapy visits at Children's Hospitals and Clinics of MN
  * Received PT evaluation within 6 months of starting cancer treatment.

Exclusion Criteria:

* • Neurological impairments prior to cancer diagnosis

  * Developmental disorders (Downs syndrome, chromosomal disorders)
  * Non-English speaking parent/child
  * Lower extremity or pelvic surgery

Ages: 7 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Diagnosed with a non-CNS cancer diagnosis with chemotherapy regimen including vincristine, carboplatin, or cisplatin greater than 5 years off of cancer treatment
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2012-12-18 (Actual); Primary Completion 2021-12-13 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Ankle range of motion | One day study
  Active and passive ankle range of motion measured by goniometry
Ankle strength | One day study
  Ankle plantarflexion and dorsiflexion dynamometry and manual muscle testing of ankle dorsiflexion and great toe extension

SECONDARY OUTCOMES:
Chemotherapy-induced peripheral neuropathy | One day study
  CIPN measured by the Pediatric Modified Total Neuropathy Scale. Scores range from 0 - 32 with higher scores correlating to greater severity in neuropathy. Cut-off score for clinical neuropathy is 4.
Foot posture | One day study
  Standing hindfoot alignment
Gait capacity | One day study
  6-minute walk test
Gait | One day study
  Spatiotemporal parameters of gait measured by Gaitrite system
Running speed | One day study
  Presidential fitness shuttle run
Balance | One day study
  Bruininks-Oseretsky Test of Motor Proficiency balance subtest
Faces pain scale and visual analog scale | One day study
  Faces pain scale and visual analog scale with scores ranging from 0-10 with higher numbers indicating greater pain level.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Minnesota, Minneapolis, Minnesota, United States